CLINICAL TRIAL: NCT03669692
Title: Open Randomized Clinical Trial to Evaluate the Effects of Intermittent Caloric Restriction in Patients With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients available
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, José Luis Ponce Díaz-Reixa, Urologist, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO - CHUAC - 002 - HBP - RC
Record Dates: First submitted 2018-09-09; First posted 2018-09-13 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Prostatic Hyperplasia, Benign; Metabolic Syndrome
Keywords: Prostate; Caloric Restriction; Metabolic Syndrome; Heart Rate Variability
MeSH Terms: conditions — Prostatic Hyperplasia; Metabolic Syndrome | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Open Randomized Clinical Trials
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients in the control group will be assigned to a free diet (ad libitum), according to the Spanish Association of Urology lifestyle recommendations for patients with LUTS
  Interventions: Behavioral: Control
- Caloric Restriction (Experimental): Patients in the experimental group will be assigned to intermittent caloric restriction, based on an early time restricted eating, with a 16/8 fasting/feeding scheme.
  The patients in this group will have a RC progressive scheme until achieve a maximum of 5 days a week of fasting.
  Interventions: Behavioral: Caloric Restriction

INTERVENTIONS:
Behavioral: Caloric Restriction — Subjects will be trained to perform intermittent caloric restriction, based on an early time restricted feeding, with a 16/8 hour fasting / feeding schedule, respectively.
  Arms: Caloric Restriction
Behavioral: Control — Subjects will receive diet and lifestyle recommendations from the Spanish Association of Urology, for symptoms secondary to HBP, without restriction in the meal schedule.
  Arms: Control

SUMMARY:
Lower urinary tract symptoms (LUTS) include filling, emptying or post-voiding state alterations; producing symptomatology depending of the underline mechanism. Benign prostatic hyperplasia (BPH) is the most common underlying disease, which increases with age and significantly affects men over 50 years. There are currently no prevention or curative treatment guidelines, as their pathophysiological mechanism is not exactly known. Several factors have been implicated, such as hormones, aging, lifestyle or diet.

BPH is associated with metabolic disorders, the basis of which is insulin resistance and its associated pathologies: diabetes, hypertension, obesity, dyslipidemia and metabolic syndrome. Patients without these metabolic signs have a lower incidence of BPH and / or LUTS. Insulin resistance (IR) is associated with greater proliferation and a reduction of cellular apoptosis at the prostate level; leading to an increase in prostate volume or symptoms. Likewise, the autonomic nervous system (ANS) imbalance, both in favor of sympathetic (emptying symptoms) or parasympathetic (filling symptoms), influences LUTS. SNA activity can be measured non-invasively, repetitively and effectively by measuring the heart rate variability (HRV).

Caloric restriction with optimal nutrition (CRON, hereinafter only CR) is the most physiologically adapted nutritional alternative to our ancestral needs and has been shown in humans to reduce insulin resistance and associated pathologies. It has also been observed that CR improves the balance of the SNA and allows to improve LUTS.

Proliferation inhibition and prostatic apoptosis induction, mediated through CR, by insulin-IGF-1 axis reduction and mTOR metabolic pathways inhibition, are the central axis of this project. CR will be used to reduce insulin resistance, IGF expression and inhibition of the PI3K / AKT / mTOR pathway, to reduce prostate cell proliferation and promote prostatic tissue apoptosis; in this way it will be possible to reduce its volume and improve the symptomatology.

Additionally, CR will allow us to evaluate the potential benefits it has on certain metabolic diseases (diabetes, dyslipidemia, obesity, hypertension, etc.), anthropometric values (BMI, abdominal perimeter and skin folds) and autonomic nervous system functionality (HRV) .

ELIGIBILITY:
Inclusion Criteria:

* Signature of specific informed consent for this study.
* Metabolic syndrome according to WHO criteria
* Current intake food pattern > 14 hours of duration.
* Total PSA below 2,5 ng/mL or total PSA 4 - 10 ng/mL and free/total PSA > 25%
* IPSS score > 9 points
* Maximal flow rate < 15 cc/secs
* Prostatic volume > 40 cc.

Exclusion Criteria:

* Active oncological disease; includes patients already treated without complete remission or in current active treatment.
* PSA 4 - 10 ng/mL and free/total PSA < 25% or PSA > 10 ng/mL
* Previous prostatic biopsy in the last 5 years.
* Treatment with prostatic phytotherapy in the last 4 weeks.
* BPH alphablocking treatment in the last 6 weeks.
* 5-alpha-reductase treatment in the last 6 months.
* Anticholinergic or betamimetics treatment in the last 4 weeks
* Eating, weight management disorder or previous bariatric surgery.
* Concurrent treatment with the following drugs in the fasting period: AAS and NSAIDs (except paracetamol).
* Concurrent treatment with any of the following steroids: prednisolone, budesonide, dexamethasone, fluidcortisone, hydrocortisone or prednisone.
* Major mental illness, which does not allow informed consent.
* Previous cardiovascular event in the last 12 months.
* Liver, gastrointestinal, renal or severe previous endocrine or decompensated disease in the last 12 months.
* Presence of significant vesical lithiasis.
* Type I diabetic patients
* Type II diabetic patients in treatment with sulfonylureas and sodium-glucose cotransport inhibitors, as well as in patients with insulin therapy.
* Loss of patient follow-up
* Non-compliance with protocol procedures.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the International Prostatic Symptoms Score (IPPS) | Change from Baseline IPPS at 36 months
  IPSS is a 7 items questionnaire (0-35 points) with 5 answers each, which analyzes the lower urinary tract symptoms. Higher scores indicate greater symptomatology. It is classified as mild up to 7 points, moderate 8-19 and severe greater than 20 points.

SECONDARY OUTCOMES:
Change in Prostatic volumen | Change from Baseline Prostatic Volumen at 36 months
  To evaluate prostatic volumen reduction, trough transrectal sonography
Change in Insulin Resistance | Change from Baseline Insulin Resistance at 36 months
  To evaluate variations on insuline resistance through the HOMA-IR formula.
Prostatic Specific Antigen (PSA) | Before and after 36 months
  To evaluate PSA variation
Testosterone | Before and after 36 months
  To evaluate Testosterone variation
IIEF5 | Before and after 36 months
  To evaluate the International Index of Erectile Function variation
Prostate Cancer | 36 months
  To evaluate prostate cancer incidence
Change in SF36 score | Change from Baseline SF36 questionnaire at 36 months
  To evaluate quality of life through SF36 questionnaire.
Tamsulosin prescription | Before and after 36 months
  To assess the incidence of the prescription of Tamsulosin for symptoms relief. It will be analyzed as a percentage of patients with Tamsulosin prescription.
Dutasteride/Finasteride prescription percentage | Before and after 36 months
  To assess the incidence of the prescription of Dutasteride or Finasteride for symptoms relief . It will be analyzed as a percentage of patients with Dutasteride or Finasteride prescription.
Surgery for BPH | Before and after 36 months
  To assess the surgical treatment needs for BPH. It will be analyzed as a percentage of patients who are operated on by TURP or simple prostatectomy.
Change in Body Mass Index (BMI) variation | Change from Baseline BMI at 36 months
  To evaluate variations on body mass index, measured as weight (kilograms) divided by height (cm) square.
Change in Abdominal perimeter variation | Change from Baseline abdominal perimeter variation at 36 months
  To evaluate variations on abdominal perimeter, measured as centimeters.
Diastolic pressure variation | Before and after 36 months
  To evaluate variations on diastolic pressure variation, measured as mmHg.
Sistolic pressure variation | Before and after 36 months
  To evaluate variations on sistolic pressure variation, measured as mmHg.
Heart rate variation | Before and after 36 months
  To evaluate variations on heart rate, measured as beats per minute.
Total cholesterol variation | Before and after 36 months
  To evaluate variations on total cholesterol, measured as mg/dL.
High Density Lipoprotein cholesterol variation | Before and after 36 months
  To evaluate variations on HDL cholesterol, measured as mg/dL.
LDL cholesterol variation | Before and after 36 months
  To evaluate variations on LDL cholesterol, measured as mg/dL.
Triglyceride variation | Before and after 36 months
  To evaluate variations on triglyceride, measured as mg/dL.
Alanine transaminase (ALT) variation | Before and after 36 months
  To evaluate variations on alanine transaminase, measured as IU.
Aspartate transaminase (AST) variation | Before and after 36 months
  To evaluate variations on aspartate transaminase, measured as IU.
HRV parameter - Parasympathetic Nervous System Index (PNS index) | Before and after 36 months
  To evaluate variations on PNS index, measured by heart rate variability, through Kubios software version 3.1. PNS index includes the following measures: Mean RR, RMSSD and high frequency (HF) power
HRV parameter - Sympathetic Nervous System Index (SNS index) | Before and after 36 months
  To evaluate variations on SNS index, measured by heart rate variability, through Kubios software version 3.1. The SNS index includes the following measures: Mean HR, Stress index and low frequency (LF) power.
HRV parameter - Low frequency / High Frequency Ratio (LF/HF ratio) | Before and after 36 months
  To evaluate variations on LF/HF ratio, measured by heart rate variability, through Kubios software version 3.1. Values upper 1.6 indicates SNS predominance.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Luis Ponce Diaz-Reixa, A Coruña, Spain